CLINICAL TRIAL: NCT02235623
Title: Randomized Trial of One Stage vs Two Stage Orchidopexy for Abdominal Undescended Testis
Brief Title: Orchidopexy Randomized Clinical Assessment
Acronym: ORCA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Caleb Nelson, Caleb Nelson, MD MPH, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00008033
Record Dates: First submitted 2014-09-02; First posted 2014-09-10 (Estimated); Last update posted 2025-01-22 (Actual); Status verified 2024-02

CONDITIONS: Unilateral Cryptorchidism
Keywords: Laparoscopic Surgery; Orchiopexy
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Stage 1- Single-stage Fowler-Stephens orchidopexy (FSO) (Other): Stage 1 single surgery to clip the vessels to the testis, divide the spermatic vessels and bring the testis into the scrotum.
  Interventions: Procedure: Single-stage Fowler-Stephens orchidopexy (FSO)
- Stage 2- Two-stage Fowler-Stephens orchidopexy (FSO) (Other): Stage 2 2 surgeries: 1st surgery-Clip vessels to testis. 2nd surgery done 6-12 months later, divide the spermatic vessels and bring the testis into the scrotum.
  Interventions: Procedure: Two-stage Fowler-Stephens orchidopexy (FSO)

INTERVENTIONS:
Procedure: Single-stage Fowler-Stephens orchidopexy (FSO)
  Arms: Stage 1- Single-stage Fowler-Stephens orchidopexy (FSO)
Procedure: Two-stage Fowler-Stephens orchidopexy (FSO)
  Arms: Stage 2- Two-stage Fowler-Stephens orchidopexy (FSO)

SUMMARY:
This is a randomized trial designed to evaluate testicular outcomes after a single stage versus a two-stage surgical procedure to fix an undescended, one-sided testicle located in the abdomen. Also to determine and compare the costs, surgical complications and the health related quality of life for the two procedures. Testicular outcomes will be measured using a scrotal ultrasound 6-12 months after the procedure (after the second stage procedure for those randomized to a 2 stage surgery).

ELIGIBILITY:
Inclusion Criteria:

* Boys age 4 months to 36 months
* Undergoing diagnostic laparoscopy for unilateral non-palpable testis, who are found at laparoscopy to have an abdominal undescended testis, in whom a Fowler-Stephens Orchiopexy would be appropriate.

Exclusion Criteria:

* Age > 36 months
* Age < 4 months
* Bilateral cryptorchidism
* Solitary testis
* Findings at laparoscopy for which Fowler-Stephens Orchiopexy would not be indicated
* Intra-operative mobility of the intra-abdominal testis such that, with no (or minimal) mobilization, the testis is able to reach the contralateral internal ring, without dividing the spermatic vessels.
* Assessment of whether a single stage primary orchidopexy will be performed, is entirely at the discretion of the attending surgeon.

Ages: 4 Months to 36 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2014-08; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the volume of the operated testis via ultrasound measurements. | 6-12 months after final FSO surgery
  To evaluate the volume of the operated testis at 6-12 months after single-stage Fowler-Stephens orchidopexy (FSO) (6-12 months after two- stage FSO), as determined by ultrasound measurements. This will be compared to the intra-operative testicular measurements done during the laparoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Caleb P Nelson, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No